CLINICAL TRIAL: NCT05583110
Title: Single Arm Phase II Study of the Efficacy and Safety of the Combination of Trastuzumab Plus TUCAtinib Plus viNorelbine in Patients With HER2-positive Non-resectable Locally Advanced or Metastatic Breast Cancer "TrasTUCAN Study"
Brief Title: Efficacy and Safety of the Combination of Trastuzumab Plus TUCAtinib Plus viNorelbine in Patients With HER2-positive Non-resectable Locally Advanced or Metastatic Breast Cancer
Acronym: TrasTUCAN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was closed early due to safety concerns and an unfavorable benefit-risk balance. Unexpected high neutropenia rates required a costly sub-study, which was not feasible, forcing the sponsor to terminate the trial prematurely.
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM/2020-08; 2021-002561-18 (EudraCT Number)
Record Dates: First submitted 2022-10-11; First posted 2022-10-17 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: HER2-positive Metastatic Breast Cancer; Locally Advanced HER2 Positive Breast Carcinoma
Keywords: tucatinib; Non-resectable locally advanced or metastatic breast cancer; HER2-positive
MeSH Terms: conditions — Breast Neoplasms | interventions — tucatinib; Trastuzumab; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trastuzumab-Vinorelbine-Tucatinib (Experimental): Trastuzumab-Vinorelbine-Tucatinib
  Interventions: Drug: Tucatinib; Drug: Trastuzumab; Drug: Vinorelbine

INTERVENTIONS:
Drug: Tucatinib — Run-in Phase:
  * Trastuzumab either IV or SC: 8 mg/kg IV loading dose (if necessary), followed by 6 mg/kg intravenous (IV) or 600 mg subcutaneous (SC) every 3 weeks.
  * Oral vinorelbine: 50 mg/m2 (in the first cycle) and 60 mg/m2 (in the following cycles if no dose limiting toxicity [DLT] is seen) on days 1 and 8, every 3 weeks.
  * Oral tucatinib 300 mg twice a day (BID) on a continuous dosing schedule.
  Following patients in the phase II:
  * Trastuzumab either IV or SC: 8 mg/kg IV loading dose (if necessary), followed by 6 mg/kg IV or 600 mg SC every 3 weeks.
  * Oral vinorelbine: 50 mg/m2 or 60 mg/m2 (based on the run-in phase results) on days 1 and 8, every 3 weeks.
  * Oral tucatinib 300 mg BID on a continuous dosing schedule.
  Other Names: Tukysa
Drug: Trastuzumab — Run-in Phase:
  * Trastuzumab either IV or SC: 8 mg/kg IV loading dose (if necessary), followed by 6 mg/kg intravenous (IV) or 600 mg subcutaneous (SC) every 3 weeks.
  * Oral vinorelbine: 50 mg/m2 (in the first cycle) and 60 mg/m2 (in the following cycles if no dose limiting toxicity [DLT] is seen) on days 1 and 8, every 3 weeks.
  * Oral tucatinib 300 mg twice a day (BID) on a continuous dosing schedule.
  Following patients in the phase II:
  * Trastuzumab either IV or SC: 8 mg/kg IV loading dose (if necessary), followed by 6 mg/kg IV or 600 mg SC every 3 weeks.
  * Oral vinorelbine: 50 mg/m2 or 60 mg/m2 (based on the run-in phase results) on days 1 and 8, every 3 weeks.
  * Oral tucatinib 300 mg BID on a continuous dosing schedule.
  Other Names: Herceptin
Drug: Vinorelbine — Run-in Phase:
  * Trastuzumab either IV or SC: 8 mg/kg IV loading dose (if necessary), followed by 6 mg/kg intravenous (IV) or 600 mg subcutaneous (SC) every 3 weeks.
  * Oral vinorelbine: 50 mg/m2 (in the first cycle) and 60 mg/m2 (in the following cycles if no dose limiting toxicity [DLT] is seen) on days 1 and 8, every 3 weeks.
  * Oral tucatinib 300 mg twice a day (BID) on a continuous dosing schedule.
  Following patients in the phase II:
  * Trastuzumab either IV or SC: 8 mg/kg IV loading dose (if necessary), followed by 6 mg/kg IV or 600 mg SC every 3 weeks.
  * Oral vinorelbine: 50 mg/m2 or 60 mg/m2 (based on the run-in phase results) on days 1 and 8, every 3 weeks.
  * Oral tucatinib 300 mg BID on a continuous dosing schedule.
  Other Names: Navelbine

SUMMARY:
Breast cancer (BC) is the most common neoplasm in the world. In Spain, one in 8 women is diagnosed with BC. The human epidermal growth factor receptor 2 (HER2)-positive BC subtype (that represents around 20% of all BC) was associated with poor prognosis however, new therapeutic advances have significantly increased the cure rate of patients in early stages.

In the metastatic setting, anti-HER2 targeted therapies have significantly improved overall survival (OS) with good quality of life, however there is still a substantial group of patients who die, and therefore additional drugs need to be investigated.

Trastuzumab, an anti HER2 antibody has demonstrated, in combination with chemotherapy, an improvement of OS in early and metastatic stages.

Tucatinib is an oral selective inhibitor of the HER2 receptor tyrosine kinase subunit. Its high affinity for this subunit causes fewer toxicities, such as rash and diarrhea, which are common with other anti-HER tyrosine kinase inhibitors (TKIs).

Vinorelbine has been evaluated previously in combination with trastuzumab showing interesting results.

This is a single country, multicenter, single arm phase II clinical trial with a safety run-in phase, to study the efficacy, safety and tolerability of the administration of tucatinib in combination with trastuzumab and vinorelbine in HER2-positive non-resectable locally advanced or metastatic breast cancer (MBC) with measurable disease.

DETAILED DESCRIPTION:
Patients with brain metastasis are allowed (but up to maximum of 50% of included patients).

Forty-nine patients will be enrolled in the study:

* The first 3 patients included in the study will receive trastuzumab plus tucatinib plus oral vinorelbine at a dose of 50 mg/m2 in the first cycle. If not dose limiting toxicity (DLT) is observed, these patients will receive oral vinorelbine at a dose of 60 mg/m2 for the following cycles.
* If 1/3 patients experience DLT in the first cycle, 3 additional patients will be included to receive trastuzumab plus tucatinib plus oral vinorelbine at a dose of 50 mg/m2 in the first cycle and then 60 mg/m2.
* If 0/3 or <2/6 patients experience DLT in the first cycle the vinorelbine dose will be 60 mg/m2 for all the following patients included in the study.
* If ≥2 out of 3 or 6 patients experienced DLT in the first cycle, all the following included patients will receive oral vinorelbine at a dose of 50 mg/m2.

DLTs are defined according to the National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 as any of the following events considered by the investigator to be related to investigational treatment:

* Grade 4 neutropenia lasting more than 7 consecutive days or associated with fever.
* Grade 4 thrombocytopenia lasting more than 7 consecutive days.
* Grade 3 thrombocytopenia associated with clinically significant bleeding.
* Platelet count <10,000/mm3.
* Delay of more than 7 days in the initiation of a subsequent cycle due to treatment-related adverse events.
* Any grade 3 or higher non-hematologic toxicity (except grade 3 or higher nausea/emesis or diarrhea in the absence of optimal symptomatic treatment for these conditions, grade 3 or higher fatigue lasting less than 1 week and other grade 3 or higher non-hematologic toxicity that could be controlled to grade 2 or less with appropriate treatment).

Justification of Sample size determination:

The A'Hern one stage design will be used for this study. Taking into account the HERCLIMB study, we assume a null hypothesis (H0) of an Objective response rate (ORR) of 23% and alternative hypothesis (H1) of an ORR of 40%. With an alpha error of 0.05 and a statistical power of 80%, we will need to include 46 evaluable patients. Assuming a 5% dropout rate, 49 patients will be included in this study.

Patients included in the run-in phase will be considered for the efficacy analysis of the phase II.

Study Duration:

The start date of the study is the date of the first site activation. Recruitment period will occur during approximately 18 months from the first patient in.

The end date of the study is the date of the last visit of the last patient (LPLV), including follow-up. The duration of the study will be approximately 40 months from the first patient in.

Performing exploratory objectives will be independent of the date of the end of the study.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be enrolled in the study only if they meet all of the following criteria:

1. Written and signed informed consent obtained prior to any study-specific procedure.
2. Male or female patients at least 18 years of age.
3. Availability of pre-treatment archival Formalin-Fixed Paraffin-Embedded (FFPE) tumor tissue (preferably the most recent available), otherwise possibility to perform a biopsy, to carry out exploratory biomarker analyses.
4. Documented HER2-positive status by local laboratory determination, preferably on the most recent available FFPE tumor sample, according to the American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) international guidelines valid at the time of the assay.
5. Previous therapy with at least two prior anti-HER2 treatment regimens (either in early stage or advanced disease). Prior taxanes and trastuzumab are mandatory. Prior treatment with pertuzumab, T-DM1, trastuzumab-deruxtecan and anti-HER2 TKI agents is allowed.
6. Measurable disease according to RECIST 1.1 criteria, defined as at least 1 extra-osseous lesion that can be accurately measured in at least 1 dimension.
7. Mandatory contrast brain magnetic resonance imaging (MRI) must be performed at baseline and patients must have at least one of the following:

   1. No evidence of brain metastases.
   2. Untreated brain metastases not needing immediate local therapy.
   3. Previously treated brain metastases.

      * Brain metastases previously treated with local therapy may either be stable since treatment or may have progressed since prior local central nervous system (CNS) therapy, provided that there is no clinical indication for immediate re-treatment with local therapy.
      * Subjects treated with CNS local therapy for newly identified lesions may be eligible to enroll if all of the following criteria are met:

        * Time since stereotactic radiosurgery (SRS) is at least 1 week prior to first dose of study treatment, time since whole brain radiation therapy (WBRT) is at least 3 weeks prior to first dose, or time since surgical resection is at least 4 weeks.
        * Other sites of evaluable disease are present.
      * Relevant records of any CNS treatment must be available to allow for classification of target and non-target lesions.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1.
9. Life expectancy ≥ 12 weeks.
10. Adequate organ and marrow function defined as follows:

    1. Absolute Neutrophil Count (ANC) ≥ 1,500/mm3 (1.5x109/L).
    2. Platelet count ≥ 100,000/mm3 (100x109/L).
    3. Hemoglobin ≥ 9g/dL (90g/L).
    4. Serum creatinine ≤ 1,5x upper limit of the normal range (ULN) or estimated creatinine clearance ≥ 60 mL/min as calculated using the standard method for the institution.
    5. Total serum bilirubin ≤ 1,5 x ULN (≤ 3.0 x ULN if Gilbert´s disease).
    6. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT ≤ 3.0 x ULN (≤5.0 x ULN if liver metastases are present).
    7. Alkaline phosphatase ≤ 2.5 x ULN (≤5.0 x ULN if bone or liver metastases are present).
11. Left ventricular ejection fraction (LVEF) ≥ 50% measured by multiple-gated acquisition scan (MUGA) or echocardiogram (ECHO).
12. Negative urine or serum pregnancy test for females of childbearing potential.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

1. Have received more than 4 lines of systemic therapy for locally advanced or MBC.
2. Have received prior treatment with tucatinib, vinorelbine for locally advanced or MBC or anti-HER2 TKI agents if administered less than 12 months prior to study entry.
3. Have used a strong CYP3A4 or CYP2C8 inhibitor or CYP3A substrate within 2 weeks, or a strong CYP3A4 or CYP2C8 inducer within 5 days prior to the first dose of study treatment (see Protocol Attachment 2 for more information).
4. Require therapy with warfarin or other coumarin derivatives (non-coumarin anticoagulants are allowed).
5. Patients who received before inclusion:

   1. Any investigational agent within 4 weeks.
   2. Chemotherapy within a period of time that is shorter than the cycle duration used for that treatment (e.g. < 3 weeks for fluorouracil, doxorubicine, epirubicin or < 1 week for weekly chemotherapy).
   3. Biologic therapy (e.g., antibodies): up to 4 weeks prior to starting study treatment.
   4. Endocrine therapy: tamoxifen or aromatase inhibitor (AI) within 2 weeks prior to starting study treatment.
   5. Corticosteroids within 2 weeks prior to starting study treatment. Note: the following uses of corticosteroids are permitted at any time: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular).
   6. Radiotherapy within 2 weeks (3 weeks if WBRT) prior to starting study treatment (all acute toxic effects must be resolved to NCI-CTCAE version 5.0 grade <1, except toxicities not considered a safety risk for the patient at investigator´s discretion). Patients who received prior radiotherapy to >25% of bone marrow are not eligible regardless of when it was administered.
   7. Major surgery or other anti-cancer therapy not previously specified within 4 weeks prior to starting study treatment, Resolution of all acute toxic effects of prior anti-cancer therapy or surgical procedures to NCI-CTCAE version 5.0 grade ≤ 1 (except alopecia or other toxicities not considered a safety risk for the patient at investigator´s discretion) is mandatory.
6. Are unable for any reason to undergo MRI of the brain.
7. Have any of the following with regards to CNS disease:

   1. Any untreated brain lesions >2 cm in size.
   2. Any brain lesion thought to require immediate local therapy, including (but not limited to) a lesion in an anatomic site where increase in size or possible treatment-related edema may pose risk to patient (e.g. brain stem lesions). Patients who undergo local treatment for such lesions identified by screening contrast brain MRI may still be eligible for the study based on criteria described under CNS inclusion criteria 7b.
   3. Known or concurrent leptomeningeal disease as documented by the investigator.
   4. Ongoing use of corticosteroids for control of symptoms of brain metastases at a total daily dose of >2 mg of dexamethasone (or equivalent).
   5. Poorly controlled (> 1/week) generalized or complex partial seizures or manifest neurologic progression due to brain metastases notwithstanding CNS-directed therapy.
8. Have clinically significant, uncontrolled heart disease and/or recent cardiac events including any of the following:

   1. Ventricular arrhythmia requiring therapy.
   2. Myocardial infarction or unstable angina within 6 months prior to first dose of study treatment.
   3. Uncontrolled hypertension (defined as persistent systolic blood pressure > 150 mm Hg and/or diastolic blood pressure > 100 mm Hg on antihypertensive medications).
   4. Any history of symptomatic congestive heart failure (CHF).
   5. History of LVEF decline below 50% during or after prior trastuzumab therapy or other cardiac toxicity during previous trastuzumab treatment that necessitated discontinuation of trastuzumab.
9. Have a diagnosis of any other malignancy within 3 years prior to inclusion, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix or colorectal.
10. Have history of allergic reactions to trastuzumab, vinorelbine, or tucatinib (or compounds chemically or biologically similar), except for Grade 1 or 2 infusion related reactions to trastuzumab or vinorelbine that were successfully managed.
11. Have difficulties to swallow tablets, malabsorption syndrome, disease significantly affecting gastrointestinal function, resection of the stomach or small bowel, or active inflammatory bowel disease (e.g., ulcerative diseases).
12. Have positive serology for Human Immunodeficiency Virus (HIV), or active infection for hepatitis B, hepatitis C or have other known chronic liver disease.
13. Other severe acute or chronic medical (such as neuropathy grade 3-4) or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
14. Are pregnant, breastfeeding, or planning a pregnancy. Women of child-bearing potential or partners of women of child-bearing potential, unless agreement to remain abstinent or use of single or combined non-hormonal contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 7 months after the last dose of study treatment.

    1. Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    2. Examples of non-hormonal contraceptive methods with a failure rate of < 1% per year include tubal ligation, male sterilization (only if he is the sole partner and have been performed at least 6 months prior to screening), and certain intrauterine devices.
    3. Alternatively, two methods (e.g., two barrier methods such as a condom and a cervical cap) may be combined to achieve a failure rate of < 1% per year. Barrier methods must always be supplemented with the use of a spermicide.
    4. Male participants must not donate sperm during study and up to the time period specified above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Approximately 26 months from the inclusion of the first patient
  Objective response rate (ORR) defined as the rate of complete response (CR) plus partial response (PR) based on the investigator's assessment using the response evaluation criteria for solid tumors (RECIST) version 1.1., out of the patients who received at least 1 dose of treatment.

SECONDARY OUTCOMES:
ORR in patients with brain metastasis at baseline | Approximately 26 months from the inclusion of the first patient
  ORR defined as the rate of complete response (CR) plus partial response (PR) based on the investigator's assessment using the response evaluation criteria for solid tumors (RECIST) version 1.1., out of the patients who received at least 1 dose of treatment in patients with brain metastasis at baseline.
Progression-free survival (PFS) | Approximately 26 months from the inclusion of the first patient
  Progression-free survival (PFS) defined as the time from the date of enrollment to the date of disease progression, based on the investigator's assessment using RECIST version 1.1., or death from any cause, whichever occurs first.
Duration of response (DOR) | Approximately 26 months from the inclusion of the first patient
  Duration of response (DOR) defined as the time from the date of first documentation of objective tumor response (CR or PR) to the date of first documented progressive disease based on the investigator's assessment using RECIST version 1.1, or death from any cause, whichever occurs first.
Disease control rate (DCR) | Approximately 26 months from the inclusion of the first patient
  Disease control rate (DCR): is defined as the rate of CR plus PR plus stable disease (SD) of any duration, based on the investigator's assessment using RECIST version 1.1 out of all enrolled patients/patients with brain metastasis.
Clinical benefit rate (CBR) | Approximately 26 months from the inclusion of the first patient
  Clinical benefit rate (CBR) defined as the rate of CR plus PR plus SD lasting more than 24 weeks, based on the investigator's assessment using RECIST version 1.1 out of all enrolled patients/patients with brain metastasis.
Overall survival (OS) | Approximately 26 months from the inclusion of the first patient
  Overall survival (OS) defined as the time from the date of enrollment to the date of death from any cause.
The Number of Participants Who Experienced Adverse Events (AE) Related to Study Treatment | Through study treatment, and average of 26 months
  Safety: Incidence and severity of AEs and clinical lab abnormalities. AE grades will be defined by the NCI-CTCAE v. 5.0. AE terms will be coded according to the MedDRA dictionary.
Change from baseline (CFB) Between Treatment Comparison in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Functional Scale Scores | Baseline, cycle 2 and 3, and then at every 2 cycles (each cycle is 21 days) and at the post-treatment visit, 30 days after last dose of study drug
  The EORTC-QLQ-C30 is a 30-item questionnaire composed of 5multi-item functional subscales (physical, role, cognitive emotional, and social functioning), 3 multi-item symptom scales (fatigue, nausea/vomiting, and pain), a global health/QoL subscale, and 6 single items assessing other cancer-related symptoms (dyspnea, sleep disturbance, appetite, diarrhea, constipation, and the financial impact of cancer). The questionnaire employs 28 4-point Likert scales with responses from "not at all" to "very much" and two 7-point Likert scales for global health and overall QoL. For functional and global QOL scales, higher scores represent a better level of functioning and are converted to a 0 to 100 scale. For symptom-oriented scales, a higher score represents more severe symptoms.
  Patients will complete EORTC QLQ-C30 at baseline, at cycle 2 and 3 and then every 2 cycles until end of treatment, and at the post-treatment visit (30 (±5) days after finishing the last dose of study drug).
Time to Deterioration (TTD) in EORTC QLQ-C30 Functional Scale | Baseline, cycle 2 and 3, and then at every 2 cycles (each cycle is 21 days) and at the post-treatment visit, 30 days after last dose of study drug
  TTD is defined as the time from the date of enrollment to the date of first detection of a deterioration event (increase of ≥ minimally important difference (MID) from baseline for the EORTC QLQ-C30 symptom scales and a decrease of ≥ MID from baseline for the EORTC QLQ-C30 functional and global health status score scales.
  The EORTC-QLQ-C30 is a 30-item questionnaire composed of 5multi-item functional subscales, 3 multi-item symptom scales, a global health/QoL subscale, and 6 single items assessing other cancer-related symptoms. The questionnaire employs 28 4-point Likert scales with responses from "not at all" to "very much" and two 7-point Likert scales for global health and overall QoL. For functional and global QOL scales, higher scores represent a better level of functioning and are converted to a 0 to 100 scale. For symptom-oriented scales, a higher score represents more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital General Universitario Gregorio Marañón, Madrid, Spain; Study Director, Study Director — Hospital Universitario Donostia, San Sebastián, Spain.; Study Director, Study Director — Hospital Universitario Reina Sofía, Córdoba, Spain
Locations (18):
- Spain (18):
  - Hospital Universitario de Jeréz De La Frontera, Cadiz, Andalusia
  - Hospital Universitario Reina Sofía, Córdoba, Andalusia
  - Hospital Universitario de Jaén, Jaén, Andalusia
  - Hospital Costa del Sol, Málaga, Andalusia
  - Hospital Universitario Virgen de Valme, Seville, Andalusia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Aragon
  - Hospital Universitario Donostia, Donostia / San Sebastian, Basque Country
  - Hospital Nuestra Señora de Sonsoles, Ávila, Castille and León
  - Hospital Clínico Universitario de Valladolid, Valladolid, Castille and León
  - ICO Badalona, Barcelona, Catalonia
  - Hospital Universitario de Bádajoz, Bádajoz, Extremadura
  - Hospital Álvaro Cunqueiro, Vigo, Galicia
  - Complejo hospitalario Universitario Insular-Materno Infantil, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital San Juan de Alicante, Alicante, Valencia
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Quironsalud Madrid, Madrid
  - Hospital Universitario de Araba, Vitoria-Gasteiz, Álava

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GEICAM is a Spanish Breast Cancer Research Group — http://www.geicam.org/